CLINICAL TRIAL: NCT03983252
Title: Effect of Alemtuzumab on Microglial Activation Assessed Using Novel [F-18]-Based Positron Emission Tomography (PET) Ligand in Multiple Sclerosis
Brief Title: Effect of Alemtuzumab on Microglial Activation Positron Emission Tomography (PET) in Multiple Sclerosis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated without recruitment.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, TARUN SINGHAL, Assistant Professor of Neurology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018A019732
Record Dates: First submitted 2019-05-31; First posted 2019-06-12 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — N-fluoroacetyl-N-(2,5-dimethoxybenzyl)-2-phenoxyaniline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relapsing Remitting Multiple Sclerosis starting Alemtuzumab (Experimental): Patients with Relapsing Remitting Multiple Sclerosis (RRMS) (defined by International Panel Criteria), age 18-60 years, enrolled to start treatment with alemtuzumab.
  Subjects will undergo [F-18]PBR06 PET scans at baseline, 6 months and 18 months.
  Interventions: Drug: [F-18]PBR06

INTERVENTIONS:
Drug: [F-18]PBR06 — PET radiopharmaceutical
  Other Names: [18F]PBR06

SUMMARY:
Specific Aims

The specific aims of the study are:

* Primary Objective: To assess the effect of alemtuzumab on microglial activation in MS patients. The hypothesis is that alemtuzumab reduces microglial activation in MS, which may mediate its effect on reducing conversion of RRMS patients to SPMS, and its effects on cognition, including cognitive fatigue.
* Secondary Objective: To determine the time course of effect of alemtuzumab on microglial activation. The hypothesis is that alemtuzumab reduces microglial activation at 6 months after initiation of treatment and this effect persists and is accentuated at 18 years, i.e. after administration of the second course

DETAILED DESCRIPTION:
I. Subject Selection

Subjects will be recruited at the Partners MS Center, 60 Fenwood Road, Boston, MA. In addition, referrals for the study will be obtained from MS Center at University of Massachusetts Medical center, Worcester, MA. Subjects will also be recruited through Health and Clinical Research OnCall websites, and from individual physician references.

II. Study Procedures

Initial Visit:

During the first visit, subjects will be adminsitered a screening questionnaire. Subjects will review and eventually sign the consent form. They will be administered standardized questionnaires for cognitive testing and/or other co-morbidities. In addition, a blood sample will be drawn for genotype testing to identify high affinity, medium affinity and low affinity binders.

Genotype Testing Blood sample drawn on the initial screening visit will be used to obtain genomic DNA for genotyping for polymorphism within the TSPO gene on chromosome 22q13.2, using a Taqman assay. High affinity and medium affinity binders will be included in the study while the low affinity binders will be excluded from the study. The blood sample will also be assessed for serum creatinine and estimated GFR because these subjects would need to undergo intravenous gadolinium contrast administration with their 3T MRIs. Blood samples will be stored for future immunophenotyping and/or other blood assays in the future.

PET Visits:

During the PET scan visits, all women subjects of child bearing age will undergo a stat quantitative serum hCG pregnancy test and only women with a negative test will undergo the radiopharmaceutical injection.

PET imaging procedures

PET scanning session will be at BWH PET scanning facility, 75 Francis Street, Boston, MA.

For PET scanning, an intravenous (IV) catheter will be inserted into the radial antecubital or other arm or hand vein for injection of tracer. Radiopharmaceutical will be injected as a bolus (approximately 4mCi for [F-18]PBR06) followed by 5 mL of saline. At the time of imaging, the subjects will be positioned in the gantry of a PET camera. Head alignment will be made, relative to the canthomeatal line, using projected laser lines whose positions are known with respect to the slice positions of the scanner. A head support apparatus will be used to minimize head motion. Brain PET data acquisition will begin at the moment of radiotracer injection. Images will be acquired using a high-resolution PET/CT scanner.

MRI Visit(s):

All subjects will undergo a 3T Brain MRI during an MRI visit that may precede or follow the PET scan visit(s) but will be perfromed within 2 weeks of each other.

MRI imaging procedures MRI scanning session will be performed at BWH MRI facility at 60 Fenwood Road, Boston, MA. MRIs will be performed with and without intravenous gadolinium-based contrast.

Imaging Data

The following data will be collected on all subjects during scanning sessions:

During PET scanning, brain images will be acquired in 3-D mode, and dynamic acquisition scans will continue for 120 minutes. A non-diagnostic CT scan will be performed for attenuation correction of PET transmission data at the time of initiation of scanning. MRI data will be acquired as described above. T2/ FLAIR and other MRI images will be coregistered with PET images

. Non Imaging/Clinical Data

The following non-imaging/clinical data will be obtained:

Expanded Disability Status Scale (EDSS) Timed 25-feet walk (T25W) MS Functional Composite (MSFC) Minimal Assessment of Cognitive Function Scale in MS (MACFIMS) battery Symbol digit modalities test (SDMT) MSQOL-54 scale (QOL) Modified fatigue Impact Scale (MFIS) Pittsburgh Sleep Quality Index (PSQI) Beck's Depression Inventory (BDI) Center for Epidemiological Studies-Depression Scale (CES-D) Hospital Anxiety and Depression Scale (HADS)

ELIGIBILITY:
Inclusion Criteria:

* Patients with Relapsing Remitting Multiple Sclerosis (RRMS) (defined by International Panel Criteria)
* Age 18-60 years
* Enrolled to start treatment with alemtuzumab

Exclusion Criteria:

* Relapse/Corticosteroid treatment in the past 4 weeks to avoid transient effects on imaging
* Individuals with a known alternate neurologic disorder, previous head injury, or substance abuse.
* Individuals with bipolar disease and schizophrenia
* Concurrent medical conditions that contraindicate study procedures.
* Women who are pregnant or nursing. Also, any woman who is seeking to become pregnant or suspects she is pregnant will be excluded from enrollment.
* Claustrophobia
* Non-MRI compatible implanted devices
* Low affinity binder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
PET Uptake/Standardized uptake value ratio (SUVR) change | baseline and 18 months
  PET outcome measure change at 18 months from baseline

SECONDARY OUTCOMES:
PET Uptake/Standardized uptake value ratio (SUVR) change | baseline and 6 months
  PET outcome measure change at 6 months from baseline
T2/FLAIR lesion load change | baseline and 18 months
  MRI outcome measure change at 18 months from baseline
Whole brain/deep gray matter atrophy change | baseline and 18 months
  MRI outcome measure change at 18 months from baseline
Expanded Disability Status Scale (EDSS) change | baseline and 18 months
  Clinical outcome measure change at 18 months from baseline; Scale Range: 0-10; Higher values represent worse outcomes
Timed 25-foot walk (T25FW) change | baseline and 18 months
  Clinical outcome measure change at 18 months from baseline
Modified Fatigue Impact Scale (MIFS) change | baseline and 18 months
  Clinical outcome measure change at 18 months from baseline; Physical subscale range: 0-36; Cognitive subscale range: 0-40; Psychosocial subscale range: 0-8; Total MFIS Score scale range (Subscales Summed): 0-84; Higher values represent worse outcomes
Minimal Assessment of Cognitive Function in MS (MACFIMS) change | baseline and 18 months
  Clinical outcome measure change at 18 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Singhal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Partners MS Center, 60 Fenwood Road, Boston, Massachusetts, United States